CLINICAL TRIAL: NCT01440647
Title: Nasal Intermittent Positive Pressure Ventilation Allows Early Extubation In Infants Less Than 28 Weeks Gestation: A Pilot Study
Brief Title: Study of Nasal Ventilation In Preterm Infants To Decrease Time on The Respirator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Olga Sorina, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-0090
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-02

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Respiration, Artificial; Infant, Premature; Bronchopulmonary Dysplasia; Continuous Positive Airway Pressure; Non-Invasive Positive-Pressure Ventilation; Intermittent Positive-Pressure Ventilation; High-Frequency Ventilation
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Aspiration; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIPPV (Experimental): Extubation to NIPPV (nasal intermittent positive pressure ventilation)
  Interventions: Procedure: Extubation to NIPPV
- CPAP (Active Comparator): After extubation this arm was placed on CPAP (continuous positive airway pressure) and was not offered NIPPV in the first month on life
  Interventions: Procedure: Extubation to CPAP

INTERVENTIONS:
Procedure: Extubation to NIPPV — After extubation infants were placed on NIPPV as soon as all the extubation criteria were met
  Other Names: NIPPV
  Arms: NIPPV
Procedure: Extubation to CPAP — After extubation infants were placed on CPAP
  Other Names: CPAP
  Arms: CPAP

SUMMARY:
Very premature infants often cannot breathe on their own and require assistance with a respirator. Conventional respirators deliver air or oxygen via a breathing tube placed through the mouth to the airway (endotracheal tube). A prolonged use of an endotracheal tube is associated with injury to the lungs. Currently, a premature baby has to be ventilated through an endotracheal tube until he/she can fully breathe independently. In the current study, in order to shorten the time with an endotracheal tube, we utilized an alternative, less invasive ventilation procedure, nasal intermittent positive pressure ventilation (NIPPV). This procedure provides help with breathing, but requires only nasal, not endotracheal tubes. We hypothesized that NIPPV might help babies breathe, at an early stage in their recovery, when they could not breathe independently yet. Thus, by switching babies at this early stage from a regular respirator to NIPPV, we should be able to shorten the use of an injurious endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24 wks and 0 days through 27 wks and 6 days by obstetric criteria.
* Infants who are intubated for respiratory distress and received surfactant within 48 hrs of life.
* Infants whose ventilator settings are: ventilatory rate ≥ 26 breaths per minute. If the baby is on the high frequency oscillatory ventilator (HFOV) settings are MAP(mean airway pressure) ≥ 9, amplitude ≥ 2xMAP and frequency ≤ 13 Hertz.
* Infants who have never been previously extubated.

Exclusion Criteria:

* Infants enrolled in competing trials.
* Participation refused by parent/attending physician/ parent unavailable for consent.
* Infants with any major congenital abnormality.
* Postoperative patients from any surgery.
* Infants in extremis/decided upon not to receive intensive care.
* Ventilator settings lower than the intervention group.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga A DeSimone, MD, Principal Investigator — The Floating Hospital for Children at Tufts Medical Center; Abbot R Laptook, MD, Study Director — Women and Infants Hospital of RI
Locations (1):
- Women and Infants Hospital of RI, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CPAP: After extubation this arm was placed on CPAP (continuous positive airway pressure)and was not offered NIPPV in the first month on life
Period: Overall Study
Arm/Group | NIPPV | CPAP
Started | 16 | 18
Completed | 14 | 15
Not Completed | 2 | 3
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- CPAP: After extubation this arm was placed on CPAP and was not offered NIPPV in the first month on life
- Total: Total of all reporting groups
Arm/Group | NIPPV | CPAP | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 18 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: weeks]
  Gestational age in weeks | 26.1 (1.1) | 25.7 (1.1) | 25.9 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Being Intubated
Time Frame: 30 days from birth
Measure: Median (Full Range); unit: days
Groups:
- NIPPV: Extubation to NIPPV when reaching extubation criteria
- CPAP: Extubation to CPAP at the discretion of the medical team after extubation criteria were reached
Arm/Group | NIPPV | CPAP
Number analyzed (Participants) | 16 | 18
days | 12.4 [0.3 to 29.5] | 6.2 [0.5 to 30]

2. Secondary Outcome: Percentage of Participants With Reintubation
Description: Reintubation rate is a measure of the efficacy of NIPPV.
Time Frame: 0-7 days post-extubation
Measure: Number; unit: % of participants with reintubation
Arm/Group | NIPPV | CPAP
Number analyzed (Participants) | 16 | 18
% of participants with reintubation | 67 | 28

ADVERSE EVENTS:
Time Frame: Participants were followed until discharge from the hospital for an average of 100 days.
Arm/Group | NIPPV | CPAP
Serious Adverse Events (participants affected / at risk) | 2/16 | 3/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIPPV (N=16) | CPAP (N=18)
Death (General disorders) | 2 (2) | 3 (3) — Death not related to NIPPV use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes